CLINICAL TRIAL: NCT05209243
Title: Phase III Study of Stereotactic Body Radiation Therapy (SBRT) Plus Standard of Care in Castration Sensitive Oligometastatic Prostate Cancer Patients.
Brief Title: START-MET HS Prostate Cancer. : SbrT & Androgen Receptor Therapy METastatic HSPC
Acronym: START-MET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación en Oncología Radioterápica - Fundación Española de Oncología Radioterápic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GICOR-SEOR 2-21
Record Dates: First submitted 2022-01-10; First posted 2022-01-26 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer; Stereotactic Body Radiation Therapy
Keywords: SBRT; Prostate cancer; Metastatic hormonosensitive prostate cancer; Second generation hormonal treatments; Oligometastatic prostate cancer; Apalutamide; Enzalutamide; Darolutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: * Interventional arm: STANDARD OF CARE + SBRT (all metastatic lesions). ADT+ RT to the primary tumor (previously not treated) + Second generation hormonal treatment
  * Control arm: STANDARD OF CARE. ADT+ RT to the primary tumor (previously not treated) + Second generation hormonal treatment
  Patients will be stratified according to prior local treatment (yes/no) or the new imaging technique used (Choline vs PSMA PET/TC).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental): STANDARD OF CARE + SBRT (all metastatic lesions). ADT+ RT to the primary tumor (previously not treated) + Second generation hormonal treatment
  Interventions: Radiation: SBRT; Radiation: STANDARD OF CARE
- Control arm (Active Comparator): STANDARD OF CARE. ADT+ RT to the primary tumor (previously not treated) + Second generation hormonal treatment
  Interventions: Radiation: STANDARD OF CARE

INTERVENTIONS:
Radiation: SBRT — SBRT (all metastatic lesions)
  Arms: Interventional arm
Radiation: STANDARD OF CARE — ADT+ RT to the primary tumor (previously not treated) + Second generation hormonal treatment

SUMMARY:
Phase III study of stereotactic body radiation therapy (SBRT) plus standard of care in castration sensitive oligometastatic prostate cancer patients, defined as androgen deprivation therapy plus radiotherapy to the primary tumor in previously not treated patients and second generation hormonal treatments (Apalutamide/Abiraterone+Prednisone/Enzalutamide) vs androgen deprivation therapy plus radiotherapy to the primary tumor in previously not treated patients plus second generation hormonal treatments, for the treatment of oligometastatic prostate cancer.

DETAILED DESCRIPTION:
A total of 266 patients with a histological diagnosis of metastatic hormone sensitive prostate cancer, with limited disease (≤ 3 lesions based on CT and Bone Scan and ≤ 5 lesions based on Choline or PSMA PET/TC) at the diagnosis or in an oligorrecurrent stage will be included in the study. Candidates will be first screened for metastatic sites through bone scintigraphy and computerised tomography (CT) scans. Those who meet the ≤3 metastatic sites criteria will be second screened for metastatic sites based on Choline or PSMA PET/TC, which will be used to define the treatment volume of metastatic disease with SBRT/HIGRT and to confirm the oligometastatic status before the inclusion in the study.

Once included in the study, patients will be randomize (1:1) to standard of care + SBRT vs standard of care.

* Interventional arm: STANDARD OF CARE + SBRT (all metastatic lesions). ADT+ RT to the primary tumor (previously not treated) + Second generation hormonal treatment
* Control arm: STANDARD OF CARE. ADT+ RT to the primary tumor (previously not treated) + Second generation hormonal treatment

Patients will be stratified according to prior local treatment (yes/no) or the new imaging technique used (Choline vs PSMA PET/TC).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histological diagnosis of prostate cancer.
2. Castration sensitive prostate cancer patients.
3. Oligometastatic disease defined as less than or equal 3 lesions based on CT and Bone Scan and less than or equal 5 lesions based on Choline or PSMA PET/TC. Bone metastases (including the spine) or/and lymph nodes metastases.
4. Informed consent is obtained from the patient.
5. Adequate bone-marrow, liver and renal function:

   * Haemoglobin ≥10 g/dL, Leucocytes ≥ 2000/mm^3, Neutrophils ≥1500/mm^3, platelets ≥1000007mm^3
   * GOT, GPT and Total Bilirrubin ≤1.5*ULN (Upper limit of normality)
   * Creatinine ≤1.5*ULN or Creatinine Clearance ≥50 ml/min^-1

Exclusion Criteria:

1. Lack of a histological diagnosis of prostate cancer.
2. Castration resistant prostate cancer patients according to PCWG3[30].
3. Metastatic disease defined as greater than or equal 3 lesions based on CT and Bone Scan and greater than or equal 5 lesions based on Choline or PSMA PET/TC.
4. Visceral metastases.
5. Tumor stage T4 according to AJCC 8th Edition Cancer staging form.
6. Prior treatment with docetaxel, second generation hormonal treatments (Apalutamide/Abiraterone+Prednisone/Enzalutamide) or bone antiresorptive therapy.
7. Presence of symptoms or signs that are indicative of urgent surgery/radiotherapy as the first treatment for the metastases disease.
8. Lesions that require SBRT treatment that exceed critical organ tolerance limits, or do not meet the criteria for the prescription of SBRT techniques used.
9. History of another neoplastic pathology which is not a currently controlled with the exception basal cell carcinomas.
10. Presence of a cardiopathy or metabolic disorder that does not recommend the treatment with second generation hormonal treatments, or the presence of inflammatory bowel disease or other pathology that does not recommend the treatment with radiotherapy.
11. Lack of informed consent or the patient's ability to give consent.
12. Participation in other clinical trials at the time of inclusion or in the 3 previous months.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Radiological progression-free survival (rPFS) | An average of two years
  based on RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall survival | 3 years
  Defined as the time from trial randomization to the date of death from any cause. Patients not experiencing an event will be censored at the last known time they were alive.
Time to cytotoxic chemotherapy | An average of two years
  Time from trial randomization to start of first cytotoxic chemotherapy
Time to PSA progression | An average of two years
  Counted from the day of randomization to the day of either first recorded biochemical progression[30]. Patients not experiencing a biochemical failure are censored at time of last assessment
Local control | 3 years
  based on RECIST 1.1 criteria
Time to castration resistance | 3 years
  Defined as the time from trial randomization until castration resistant status
Time to skeletal-related event | An average of two years
  Time from randomization until the occurrence of a skeletal related event (SRE)
Quality of life. FACT-P | Three years after the study completion
  FACT-P
Safety profile | Three years after the study completion
  To determine acute and late toxicity due to radiotherapy, scored using the Common Terminology Criteria for Adverse Events (CTCAE) versión 4.3.
Pain. BPI | Three years after the study completion
  Evaluate the impact of the treatment on the patient's quality of life using the Brief Pain Inventory (BPI) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Antonio J Conde Moreno, MD PhD, Principal Investigator — Grupo de Investigación Clínica en Oncología Radioterápica; Fernando López Campos, MD PhD, Principal Investigator — Grupo de Investigación Clínica en Oncología Radioterápica; Alfonso Gómez-Iturriaga, MD PhD, Principal Investigator — Grupo de Investigación Clínica en Oncología Radioterápica
Locations (2):
- Spain (2):
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No